CLINICAL TRIAL: NCT02050698
Title: Hard-soled Shoe Versus Short Leg Walking Cast for a Fifth Metatarsal Avulsion Fracture: A Randomized Multicenter Noninferiority Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Hyong Nyun Kim, Professor, Hallym University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2014-OS01
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Metatarsal Fracture; Treatment
Keywords: fift metatarsal avulsion fracture; hard-soled shoe; short leg walking cast; protected weightbearing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- short leg walking cast (Active Comparator): After 1 weeks of immobilization in a short leg posterior splint, patient is allowed protected weightbearing in a short leg walking cast
  Interventions: Procedure: Protected weightbearing in a short leg walking cast
- hard-soled shoe (Experimental): After 1 weeks of immobilization in a short leg posterior splint, patient is allowed tolerable weightbearing in a hard-soled shoe
  Interventions: Procedure: Protected weightbearing in a hard-soled shoe

INTERVENTIONS:
Procedure: Protected weightbearing in a hard-soled shoe — Patients allocated to experiment group are allowed tolerable weightbearing in a hard-soled shoe after one week of immobilization in a posterior splint
  Arms: hard-soled shoe
Procedure: Protected weightbearing in a short leg walking cast — Patients allocated to control group are allowed tolerable weightbearing in a short leg walking cast after one week of immobilization in a posterior splint
  Arms: short leg walking cast

SUMMARY:
Fifth metatarsal avulsion fractures are common and can usually be treated conservatively. Symptomatic care consisting of protected weightbearing in a hard-soled shoe, air-cast walking boot, or below-knee walking cast have been successful. Several papers reported that early rehabilitation may decrease ankle stiffness, muscle and bone atrophy, and aids in early return to activities. However, early motion of the ankle joint may have the risk of displacement of the fifth metatarsal avulsion fractures. However, studies using hard-sole shoe for protected weightbearing and allowing motion of the ankle joint had successful results. Clapper et al. compared the results of hard-soled shoe and walking cast for a fifth metatarsal avulsion fracture and reported that all avulsion fractures healed uneventfully and that the results were similar between the two. However, this was not a randomized controlled trial.

Devices such as air-cast walking boot, plaster slipper, or Jone's dressing can also be used for the treatment. However, we decided to compare results of hard-soled shoe and short leg walking cast for the treatment of a fifth metatarsal avulsion fracture.

We hypothesized that the 100mm visual analogue scale (VAS) assessed on 6 months after a fifth metatarsal avulsion fracture treated with protected weightbearing in a hard-soled shoe is not inferior to protected weightbearing in a short leg walking cast but is superior to short leg walking cast with respect to time to return to normal daily life and patient's satisfaction.

DETAILED DESCRIPTION:
This study is a noninferiority, randomized controlled trial of patients presenting to multiple centers. The primary outcome measure is the 100mm VAS assessed on 6 months after a fifth metatarsal avulsion fracture. 100mm VAS was compared between the experimental group (hard-soled shoe) and the control group (short leg walking cast) on 6 months follow-up examination. The 100mm VAS is widely used self assessment tool for evaluating pain after fracture. The secondary objectives were to determine whether hard-soled shoe was superior to short leg walking cast with respect to time until return to normal daily life and patient's satisfaction.

The sample size was determined using methods appropriate for noninferiority trials, assuming 90% power and a significance level of 0.05. We performed a pilot study on 18 patients and assessed 100mm VAS on 6 months. Pooled standard deviation was 16.6. To find out whether the hard-soled shoe is not inferior to short leg walking cast for a fifth metatarsal avulsion fracture, 74 patients were required to have 90% power that the lower limit of an one-sided 95% confidence interval for the difference between two treatments will be above the noninferiority margin of -10. We assumed the drop-out rate to be 20%. Adding this number, 96 patients were required for the study.

Determination of the noninferiority margin was based on clinical significance. Todd et al. reported on a study of 48 patients that the minimum clinically significant difference of 100mm VAS was 13mm and that differences of less than this amount, even if statistically significant, are unlikely to be of clinical significance. We decided that the noninferiority margin at 10 mm difference which is less than this amount will be adequate to prove noninferiority of the experiment group (hard-soled shoe) over the control group (short leg walking cast).

After 1 weeks of immobilization in a short leg posterior splint, patients are randomized to experiment group (hard-soled shoe) and control group (short leg walking cast). Randomization was stratified by the study centers. Block randomization were used and the investigators were blinded to the block sizes being used to ensure allocation concealment. Delayed union was defined as a lack of bridging callus on 3 of 5 cortices at 12 weeks. Nonunion was defined as lack of cortical bridging or a clearly visible fracture line, at 14 weeks post injury.

If a subject had discontinued prior to completion of 6 months, the last observation was carried forward for the intent-to-treat analysis. Subjects who crossed over to the other treatment arm, for an example, patients in experiment group(hard-soled shoe) who changed to short leg walking cast or in control group (short leg walking cast) who changed to hard-soled shoe, were analyzed according to their initial group allocation for the intent-to-treat analysis. Additionally, an as-treated (per-protocal) analysis was also conducted on patients who completed the 6 months follow-up with the protocol assigned.

Although previous studied have not documented an increase risk of reduction loss with protected weightbearing in a hard-soled shoe protocol, a safety rule was put in place to assure patients, clinicians, and the health research ethics board that the safety of our patients was a priority. Reduction loss was not a primary outcome, but it was monitored carefully regardless of published evidence. A safety rule established a priori eliminated any dissent among the research team and participating surgeons about stopping the study in the event of an apparent adverse outcome related to protected weightbearing in a hard-soled shoe. If a difference of greater than three spontaneous reduction loss occurred between the groups, the intervention would be halted. A reduction loss or metal failure was defined as one that occurred without patient instigation of inappropriate activity. The reduction loss was to be monitored by study personnel not involved in the outcome assessment.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* fifth metatarsal avulsion fracture

Exclusion Criteria:

* open fractures
* pathologic fractures
* a fifth metatarsal avulsion fracture combined with other lower extremity injuries such as Lisfranc injury
* patients with diabetes or neuroarthropathy
* patients with obesity (BMI >30, weight >100 kg)
* any other conditions that are expected to prevent the patients from following the study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
100mm visual analogue scale (VAS) | 6 months after a fifth metatarsal avulsion fracture
  The 100mm VAS is widely used self assessment tool for evaluating pain after fracture.

SECONDARY OUTCOMES:
Time to return to preinjury activity | upto 6 months
patients' subjective satisfactions | 3, 5, 8, 12 weeks and 6 months after injury

CONTACTS AND LOCATIONS:
Overall Officials: Hyong Nyun Kim, MD, PhD, Study Chair — Kangnam Sacred Heart Hospital, Hallym University College of Medicine; Hyong Nyun Kim, MD, PhD, Study Director — Kangnam Sacred Heart Hospital, Hallym University College of Medicine
Locations (3):
- South Korea (3):
  - Sanbon Hospital, Wonkwang University College of Medicine, Gunpo, Gyeongi
  - CHA Bundang Medical Center, CHA University, Seongnam, Gyeongi
  - Kangnam Sacred Heart Hospital, Hallym University College of Medicine, Seoul

REFERENCES:
- [Background] Todd KH, Funk KG, Funk JP, Bonacci R. Clinical significance of reported changes in pain severity. Ann Emerg Med. 1996 Apr;27(4):485-9. doi: 10.1016/s0196-0644(96)70238-x. PMID 8604867
- [Background] Clapper MF, O'Brien TJ, Lyons PM. Fractures of the fifth metatarsal. Analysis of a fracture registry. Clin Orthop Relat Res. 1995 Jun;(315):238-41. PMID 7634674
- [Background] Gray AC, Rooney BP, Ingram R. A prospective comparison of two treatment options for tuberosity fractures of the proximal fifth metatarsal. Foot (Edinb). 2008 Sep;18(3):156-8. doi: 10.1016/j.foot.2008.02.002. Epub 2008 May 19. PMID 20307430
- [Background] Heineck J, Wolz M, Haupt C, Rammelt S, Schneiders W. Fifth metatarsal avulsion fracture: a rational basis for postoperative treatment. Arch Orthop Trauma Surg. 2009 Aug;129(8):1089-92. doi: 10.1007/s00402-008-0756-x. Epub 2008 Sep 26. PMID 18818936
- [Background] Shahid MK, Punwar S, Boulind C, Bannister G. Aircast walking boot and below-knee walking cast for avulsion fractures of the base of the fifth metatarsal: a comparative cohort study. Foot Ankle Int. 2013 Jan;34(1):75-9. doi: 10.1177/1071100712460197. PMID 23386764
- [Background] Vorlat P, Achtergael W, Haentjens P. Predictors of outcome of non-displaced fractures of the base of the fifth metatarsal. Int Orthop. 2007 Feb;31(1):5-10. doi: 10.1007/s00264-006-0116-9. Epub 2006 May 23. PMID 16721621
- [Background] Wiener BD, Linder JF, Giattini JF. Treatment of fractures of the fifth metatarsal: a prospective study. Foot Ankle Int. 1997 May;18(5):267-9. doi: 10.1177/107110079701800504. PMID 9167925